CLINICAL TRIAL: NCT05130827
Title: Pilot Trial of Plinabulin and Pegfilgrastim to Reduce the Duration of Absolute Neutropenia After Autologous Hematopoietic Cell Transplantation for Patients With Multiple Myeloma
Brief Title: Study of Plinabulin and Pegfilgrastim in People With Multiple Myeloma Undergoing an Autologous Hematopoietic Stem Cell Transplant (AHCT)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: BeyondSpring Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-337
Record Dates: First submitted 2021-11-22; First posted 2021-11-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Plinabulin; Pegfilgrastim; Autologous Hematopoietic Stem Cell Transplant (AHCT); 21-337
MeSH Terms: conditions — Multiple Myeloma | interventions — NPI 2358

STUDY DESIGN:
Intervention Model Description: This is a pilot trial investigating a single dose of plinabulin on day of stem cell infusion (Day 0) in conjunction with pegfilgrastim on Day +1 after autologous hematopoietic cell transplant (AHCT).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Plinabulin (Experimental): In this pilot study, 15 patients age 18-75 with multiple myeloma will be admitted to the hospital and treated with a single dose of high dose melphalan. Stem cell infusion will occur per institutional standard of care. Patients will then receive plinabulin 40mg flat dose IV infusion, infused over approximately 30 minutes starting between 1-3 hours after stem cell infusion on day 0. Pegfilgrastim 6mg will be administered as per standard of care on day +1.
  Interventions: Drug: Plinabulin

INTERVENTIONS:
Drug: Plinabulin — 40mg flat dose IV infusion, infused over approximately 30 minutes starting between 1-3 hours after stem cell infusion on day 0.

SUMMARY:
This study will see how long it takes for white blood cell counts to return to normal in people with multiple myeloma (MM) who receive plinabulin and pegfilgrastim after undergoing an autologous hematopoietic stem cell transplant (AHCT).

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of multiple myeloma by the enrolling institution in patient undergoing autologous HCT with melphalan 140 or 200 mg/m^2
* Age 18-75
* Have at least 3 x 10^6 CD34+ autologous stem cells/kg to be infused
* Karnofsky performance greater than or equal to 60 within 2 weeks prior to enrollment.
* Organ function testing within 28 days before enrollment:

  1. LVEF ≥45% by MUGA or rest ECHO
  2. Diffusion capacity >45% (adjusted for hemoglobin) as predicted by pulmonary function testing
* Clinical laboratory values meeting the following criteria within 14 days before enrollment:

  1. Platelet count ≥ 20 x 109/L
  2. ALT and AST ≤ 2.5 x ULN
  3. Total bilirubin ≤ 2.5 x ULN; except if the elevation is due to Gilbert's syndrome
  4. Calculated creatinine clearance > 40 mL/min
* All women of childbearing potential must:

  1. Have a negative serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) within 14 days prior to enrollment (and pre-AHCT per institutional guidelines)
  2. For 180 days after receiving plinabulin practice a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: e.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject)
  3. For 180 days after receiving plinabulin, a woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction
  4. Not of childbearing potential is defined as postmenopausal (>45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 IU/mL); permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy
  5. Note: If the childbearing potential changes after start of the study (e.g., woman who is not heterosexually active becomes active) a woman must begin a highly effective method of birth control, as described above.
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm for 180 days after receiving plinabulin

Exclusion Criteria:

* Other malignancy within the past 2 years, except for the following if treated and not active: basal cell or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or International Federation of Gynecology and Obstetrics (FIGO) Stage 1 carcinoma of the cervix
* Clinically significant infection, including known HIV or hepatitis C infection, or known hepatitis B (Hep B) surface antigen positivity. Patients with Hep B Core Antibody positivity can be enrolled if the Hep B PCR is negative, and they are on antiviral suppression.
* Patients with uncontrolled systemic fungal, bacterial, viral, or other infection despite appropriate treatment at the time of enrollment.
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 14 days or 5 half-lives before enrollment
* Had hospitalization for infection or major surgery (e.g., requiring general anesthesia) within 14 days before enrollment or have not fully recovered from surgery. Note: subjects with surgical procedures conducted under local anesthesia may participate
* A woman who is pregnant or breast-feeding, or a woman who is planning to become pregnant or a man who plans to father a child while enrolled in this study or within 180 days after plinabulin
* Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol, as judged by the PI; or unwillingness or inability to follow the procedures required in the protocol.
* Significant cardiovascular history:

  * History of myocardial infarction or ischemic heart disease within 1 year (within a window of up to 18 days less than 1 year) before study drug administration
  * Uncontrolled arrhythmia
  * History of congenital QT prolongation
  * Electrocardiogram (ECG) findings consistent with active ischemic heart disease
  * New York Heart Association Class III or IV cardiac disease;
  * Uncontrolled hypertension: blood pressure consistently >150 mm Hg systolic and > 100 mm Hg diastolic in spite of antihypertensive medication
* Prior transient ischemic attack or cerebrovascular accident with in the past year (within an 18-day window). Any neurologic toxicities ≥ Grade 2 within 3 weeks of randomization.
* History of hemorrhagic diarrhea, inflammatory bowel disease or active uncontrolled peptic ulcer disease. (Concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable). History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility.
* Known prior hypersensitivity reaction to any product containing polysorbate 80, polyoxyethylene 15-hydroxystearate/Macrogol 15 hydroxystearate (Solutol HS 15/Kolliphor HS 15).
* Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient. Examples of such conditions include uncontrolled diabetes, infection requiring parenteral anti-infective treatment, liver failure, any altered mental status or any psychiatric condition that would interfere with the understanding of the informed consent form.
* Unwilling or unable to comply with procedures required in this protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Average duration of absolute neutropenia | 1 year
  defined as the number of days after treatment in which the absolute neutrophil count is less than 500 x 10^6/L.

SECONDARY OUTCOMES:
Incidence of toxicities | 1 year
  CTCAE Version 5 will be utilized for toxicity evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Shah, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm